CLINICAL TRIAL: NCT07034300
Title: Comparison of Lidocaine Alone Versus Lidocaine With Dexmedetomidine for Intravenous Regional Anesthesia (IVRA)
Brief Title: Lidocaine vs. Lidocaine With Dexmedetomidine for Intravenous Regional Anesthesia (IVRA) in Upper Limb Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fatima Memorial Hospital (Other)
Responsible Party: Principal Investigator, Muhammad Mansoor Younas, Principal Investigator, Fatima Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMY-LidoDex-IVRA-2025
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Post-operative Pain; Upper Limb Surgery; Regional Anesthesia
Keywords: Intravenous Regional Anesthesia; Lidocaine; Dexmedetomidine; Pain; Upper Limb Surgery; Bier Block
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Lidocaine; Pharmaceutical Preparations; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Active Comparator): Intravenous Regional Anesthesia with 40 ml of 0.5% lidocaine
  Interventions: Drug: Lidocaine (drug)
- Lidocaine with Dexmedetomidine (Experimental): Intravenous Regional Anesthesia with 40 ml of 0.5% lidocaine + dexmedetomidine (0.5 μg/kg)
  Interventions: Drug: Lidocaine (drug); Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Lidocaine (drug) — 40 ml of 0.5% lidocaine
Drug: Dexmedetomidine — Dexmedetomidine (0.5 μg/kg)
  Arms: Lidocaine with Dexmedetomidine

SUMMARY:
This study compares lidocaine alone vs. lidocaine with dexmedetomidine in Intravenous regional anesthesia (IVRA) for upper limb surgery in terms of pain scores and duration of analgesia

DETAILED DESCRIPTION:
Intravenous regional anesthesia effectively anesthetizes limbs for surgeries lasting under one hour. This method involves applying a pneumatic tourniquet and injecting a local anesthetic below the tourniquet to directly target major nerves. Intravenous regional anesthesia has certain limitations, including tourniquet-related pain, risk of local anesthetic systemic toxicity, limited postoperative pain relief, and the potential risk of compartment syndrome. Despite these concerns, it remains a reliable technique with reported success rates between ninety-four percent and ninety-eight percent.

This technique, originally introduced by August Bier, isolates the limb using pressure and a pneumatic tourniquet to retain the anesthetic effect in the target area. Lidocaine, a commonly used amide-type local anesthetic, was popularized for this method after successful use in 1963. However, lidocaine alone has limitations, such as incomplete sensory nerve block, discomfort from the tourniquet, and minimal pain control after the tourniquet is released. To improve these outcomes, additives have been combined with local anesthetics to enhance pain relief after the procedure and reduce intraoperative discomfort. However, the use of such additives has been limited due to concerns about side effects or uncertain effectiveness.

Alpha-2 adrenergic receptor agonists have recently gained attention for their sedative, pain-relieving, and cardiovascular-stabilizing effects in the perioperative setting. These agents can reduce the need for general anesthesia and prolong the effects of local anesthetics in regional anesthesia techniques. Clonidine, one such medication, when added to local anesthetics, has been associated with improved pain control in spinal, epidural, and peripheral nerve blocks compared to the use of local anesthetics alone. Dexmedetomidine, a highly selective alpha-2 adrenergic receptor agonist, offers a rapid onset of action and is recognized for its beneficial sedative and pain-relieving properties.

Dexmedetomidine has additional pharmacological effects, including lowering blood pressure, reducing anxiety, and providing sedation. These properties make it useful in clinical practice, especially in the management of surgical pain and in maintaining comfort for patients in critical care settings. It is often used both during surgical procedures and for sedation in intensive care units.

Studies comparing the use of lidocaine alone versus lidocaine combined with dexmedetomidine have shown that the combination significantly improves the duration of postoperative pain relief and reduces patient-reported pain levels. One study reported a longer duration of pain relief and lower pain scores in patients who received dexmedetomidine along with lidocaine. Another study found similar improvements in both the length of pain relief and pain intensity scores when the combination was used. Despite these promising results, there is a noticeable lack of research on this topic within Pakistan, largely due to the previous unavailability of dexmedetomidine in the local market. Therefore, this study was designed to compare the effectiveness of lidocaine alone versus lidocaine combined with dexmedetomidine in the setting of intravenous regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology Status I
* American Society of Anesthesiology Status II
* Elective surgery
* Surgery duration <45 minutes

Exclusion Criteria:

* Sleep apnea
* BMI >30
* Heart block
* uncontrolled hypertension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-08-21 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Duration of Postoperative Analgesia | Up to 24 hours post surgery
  Time from surgery to first request for pain relief

SECONDARY OUTCOMES:
Pain Score according to Visual Analogue Scale (VAS) | 2 hours post-operation
  Mean Pain Score according to Visual Analogue Scale (VAS) measured on a 0-10 scale, 0 being no pain at all and 10 meaning worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad M Younas, MBBS, Principal Investigator — Fatima Memorial Hospital
Locations (1):
- Department of Anesthesiology, Fatima Memorial Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional policy and data privacy considerations. The data are not intended for secondary use beyond the scope of this study.